CLINICAL TRIAL: NCT04291768
Title: Short Course Antibiotic Treatment of Gram-negative Bacteremia: A Multicenter, Randomized, Non-blinded, Non-inferiority Interventional Study
Brief Title: Shortened Antibiotic Treatment of 5 Days in Gram-negative Bacteremia
Acronym: GNB5
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Benfield (Other)
Responsible Party: Sponsor-Investigator, Thomas Benfield, Clinical Professor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 190801; 2019-003282-17 (EudraCT Number); H-19085920 (Other: National Ethics Comittee of Denmark)
Record Dates: First submitted 2020-02-24; First posted 2020-03-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Gram-negative Bacteremia; Urinary Tract Infection Bacterial
Keywords: Gram-negative bacteremia; Urinary tract infection; Shortened antibiotic treatment; Bacterial infection
MeSH Terms: conditions — Urinary Tract Infections; Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Shortened antibiotic treatment of 5 days
  Interventions: Other: Shortened antibiotic treatment
- Control group (Active Comparator): Standard antibiotic treatment of minimum 7 days at the discretion of treating physician
  Interventions: Other: Standard antibiotic treatment

INTERVENTIONS:
Other: Shortened antibiotic treatment — Shortened antibiotic treatment of 5 days. Participation in the study will only affect treatment duration and will have no influence on the choice of treatment in respect to type and dose of antibiotic treatment.
  Arms: Intervention group
Other: Standard antibiotic treatment — Standard antibiotic treatment of minimum 7 days at the discretion of treating physician. Participation in the study will only affect treatment duration and will have no influence on the choice of treatment in respect to type and dose of antibiotic treatment.
  Arms: Control group

SUMMARY:
GNB5 is an investigator-initiated multicentre non-inferiority randomized controlled trial which aims to assess the efficacy and safety of shortened antibiotic for patients hospitalized with a Gram negative bacteremia with a urinary tract source of infection (GNB).

Five days after initiation of antimicrobial therapy for GNB, participants are randomized 1:1 to parallel treatment arms: 5 days (intervention) or minimum 7 days (control) of antibiotic treatment. The intervention group discontinues antibiotics at day 5 if clinically stable and afebrile. The control group receives antibiotics for a duration of 7 days or longer at the discretion of the treating physician.

The primary outcome is 90-day survival without clinical or microbiological failure to treatment, which will be tested with a non inferiority margin of 10%.

DETAILED DESCRIPTION:
Introduction: Prolonged use of antibiotics is closely related to antibiotic-associated infections, anti-microbial resistance and adverse drug events. The optimal duration of antibiotic treatment for Gram-negative bacteremia (GNB) with a urinary tract source of infection is poorly defined.

Methods and analysis: Investigator initiated multicenter, non-blinded, non-inferiority randomized controlled trial with two parallel treatment arms. One arm will receive shortened antibiotic treatment of 5 days and the other arm will receive standard antibiotic treatment of 7 days or longer. Randomization will occur in equal proportion (1:1) no later than day 5 of efficacious antibiotic treatment as determined by antibiogram. Immunosuppressed patients and those with GNB due to non-fermenting bacilli (Acinetobacter spp, Pseudomonas spp), Brucella spp, Fusobacterium spp or polymicrobial growth are ineligible.

Primary endpoint is 90-day survival without clinical or microbiological failure to treatment. Secondary endpoints include all-cause mortality, total duration of antibiotic treatment, hospital re-admission and Clostridioides difficile infection. Interim safety analysis will be performed after the recruitment of every 100 patients. Given an event rate of 12%, a margin of 10% and 90% power, the required sample size to determine non-inferiority is 380 patients. Analyses will be performed on both intention-to-treat and per-protocol populations.

Ethics and dissemination: Approval by Ethics Committee and National Competent Authorities will be obtained before initiation of the trial. Results of the main trial and each of the secondary endpoints will be submitted for publication in a peer-reviewed journal.

Impact: Demonstration of non-inferiority will provide needed evidence to safely shorten antibiotic treatment duration in GNB with a urinary tract source of infection and thereby reduce the risk of adverse events and development of resistance associated with use of antibiotics

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Blood culture positive for Gram-negative bacteria
* Evidence of urinary tract source of infection (positive urine culture or at least one clinical symptom compatible with urinary tract infection)
* Antibiotic treatment with antimicrobial activity to Gram-negative bacteria administrated within 12 hours of first blood culture
* Temperature <37.8°C at randomization
* Clinically stabile at randomization (systolic blood pressure > 90 mm Hg, heart rate <100 beats/min., respiratory rate <24/minute, peripheral oxygen saturation > 90 %)
* Oral and written informed consent

Exclusion Criteria:

* Antibiotic treatment (>2 day) with antimicrobial activity to Gram-negative bacteria within 14 days of inclusion
* Gram-negative bacteremia within 30 days of blood culture
* Immunosuppression (Untreated HIV-infection, Neutropenia (absolute neutrophil count < 1.0 x 109/l), Untreated terminal cancer, Receiving immunosuppressive agents (ATC-code L04A), Corticosteroid treatment (≥20 mg/day prednisone or the equivalent for >14 days) within the last 30 days, Chemotherapy within the last 30 days, Immunosuppressed after solid organ transplantation, Asplenia)
* Polymicrobial growth in blood culture
* Bacteremia with non-fermenting Gram-negative bacteria (Acinetobacter spp, Burkholderia spp, Pseudomonas spp), Brucella spp, or Fusobacterium spp
* Failure to remove source of infection within 72 hours of first blood culture (e.g. change of catheter á demeure)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
90-day survival without clinical or microbiological failure to treatment | 90 days
  90-day survival without clinical or microbiological failure to treatment as defined:
  1. All-cause mortality from day of randomization and until day 90
  2. Microbiological failure: Recurrent bacteremia due to the same microorganism as verified by sequence analysis occurring from day of randomization and until day 90
  3. Clinical failure: Re-initiation of therapy against Gram-negative bacteremia for more than 48 hours due to clinical worsening suspected to be due to the initial infecting organism and for which there is no alternate diagnosis/pathogen suspected from the day of randomization and until day 90
     1. Distant complications of initial infection, defined by growth of the same bacteria as in the initial bacteremia (e.g. endocarditis, meningitis)
     2. Local suppurative complication that was not present at infection onset (e.g. renal abscess in pyelonephritis)

SECONDARY OUTCOMES:
Mortality | 14, 30 and 90 days
  Number of deaths by any cause
Total duration of antibiotic treatment | 90 days
  Days that the participant receives antibiotic treatment for Gram-negative bacteremia, adding intravenous and oral therapy
Type of antibiotic treatment | 90 days
  Antibiotic treatment for Gram-negative bacteremia given by antibiogram
Duration of antibiotic treatment | 90 days
  Duration of antibiotic treatment for Gram-negative bacteremia given by antibiogram
Total length of hospital stay | 90 days
  Days from the date of hospital admission for Gram-negative bacteremia to the date of discharge
Hospital re-admission | 30 and 90 days
  Number of participants with readmissions for reasons related to or unrelated to Gram-negative bacteremia
Antibiotic adverse events | 90 days
  Number of participants with adverse events with possible relation to the antibiotic treatment of Gram-negative bacteremia
Use of antimicrobials after discharge | 90 days
  Days of antibiotic treatment for any reason after hospital discharge
Severe adverse events | 90 days
  Number of participants with serious adverse events according to International Council of Harmonisation-Good Clinical Practice (ICH-GCP) guidelines
Acute kidney injury | 90 days
  Number of participants with acute kidney injury is defined according to RIFLE criteria as increased creatinine level x 1.5 from baseline or estimated glomerular filtration rate (eGFR) decrease >25% or urine output of <0.5 ml/kg/h for 6 hours.
Clostridioides difficile infection | 90 days
  Number of participants with Clostridioides difficile infection
Multidrug-resistance organism | 90 days
  Multidrug-resistance organism defined as identification of resistant bacteria in a clinical specimen obtained only from a clinical infection.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Tingsgård, MD, Principal Investigator — Hvidovre University Hospital
Locations (13):
- Denmark (13):
  - University Hospital of Aalborg, Aalborg
  - University Hospital of Aarhus, Aarhus
  - Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hospital, Hellerup
  - Herlev Hospital, Herlev
  - Herning Hospital, Herning
  - Nordsjaellands Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Kolding Hospital, Kolding
  - Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
  - Regionshospitalet Silkeborg, Silkeborg

IPD SHARING:
Plan to Share IPD: Yes
Demographics, medical history, and laboratory data will be preserved to validate and replicate described research. Study protocol and statistical analysis plan will be publicly available.
  Data will be collected in the electronic data capture system (REDCap) and analyzed using open-source statistical packages in R. Data will be available immediately following the publication of the primary outcome. Data will be preserved for 10 upon study start. Anonymized trial data will be made available through relevant public databases when the trial ends. On request, anonymized patient-level data, the statistical code, and other relevant supporting information will be made available by contact with the corresponding author. Study data will be published only in pseudonymous form. Compliance with the plan will be monitored by the primary investigator routinely.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available immediately following the publication of the primary outcome. Data will be preserved for 10 upon study start.
Access Criteria: On request, anonymized patient-level data, the statistical code, and other relevant supporting information will be made available by contact with the corresponding author.

REFERENCES:
- [Background] Kang CI, Kim SH, Park WB, Lee KD, Kim HB, Kim EC, Oh MD, Choe KW. Bloodstream infections caused by antibiotic-resistant gram-negative bacilli: risk factors for mortality and impact of inappropriate initial antimicrobial therapy on outcome. Antimicrob Agents Chemother. 2005 Feb;49(2):760-6. doi: 10.1128/AAC.49.2.760-766.2005. PMID 15673761
- [Background] Biedenbach DJ, Moet GJ, Jones RN. Occurrence and antimicrobial resistance pattern comparisons among bloodstream infection isolates from the SENTRY Antimicrobial Surveillance Program (1997-2002). Diagn Microbiol Infect Dis. 2004 Sep;50(1):59-69. doi: 10.1016/j.diagmicrobio.2004.05.003. PMID 15380279
- [Background] de Kraker ME, Jarlier V, Monen JC, Heuer OE, van de Sande N, Grundmann H. The changing epidemiology of bacteraemias in Europe: trends from the European Antimicrobial Resistance Surveillance System. Clin Microbiol Infect. 2013 Sep;19(9):860-8. doi: 10.1111/1469-0691.12028. Epub 2012 Oct 8. PMID 23039210
- [Background] Sogaard M, Norgaard M, Dethlefsen C, Schonheyder HC. Temporal changes in the incidence and 30-day mortality associated with bacteremia in hospitalized patients from 1992 through 2006: a population-based cohort study. Clin Infect Dis. 2011 Jan 1;52(1):61-9. doi: 10.1093/cid/ciq069. PMID 21148521
- [Background] DANMAP 2017 - Use of antimicrobial agents and occurrence of antimicrobial resistance in bacteria from food animals, food and humans in Denmark. 2017
- [Background] Goossens H, Ferech M, Vander Stichele R, Elseviers M; ESAC Project Group. Outpatient antibiotic use in Europe and association with resistance: a cross-national database study. Lancet. 2005 Feb 12-18;365(9459):579-87. doi: 10.1016/S0140-6736(05)17907-0. PMID 15708101
- [Background] Lessa FC, Mu Y, Bamberg WM, Beldavs ZG, Dumyati GK, Dunn JR, Farley MM, Holzbauer SM, Meek JI, Phipps EC, Wilson LE, Winston LG, Cohen JA, Limbago BM, Fridkin SK, Gerding DN, McDonald LC. Burden of Clostridium difficile infection in the United States. N Engl J Med. 2015 Feb 26;372(9):825-34. doi: 10.1056/NEJMoa1408913. PMID 25714160
- [Background] Cunha BA. Antibiotic side effects. Med Clin North Am. 2001 Jan;85(1):149-85. doi: 10.1016/s0025-7125(05)70309-6. PMID 11190350
- [Background] Tamma PD, Avdic E, Li DX, Dzintars K, Cosgrove SE. Association of Adverse Events With Antibiotic Use in Hospitalized Patients. JAMA Intern Med. 2017 Sep 1;177(9):1308-1315. doi: 10.1001/jamainternmed.2017.1938. PMID 28604925
- [Background] Branch-Elliman W, O'Brien W, Strymish J, Itani K, Wyatt C, Gupta K. Association of Duration and Type of Surgical Prophylaxis With Antimicrobial-Associated Adverse Events. JAMA Surg. 2019 Jul 1;154(7):590-598. doi: 10.1001/jamasurg.2019.0569. PMID 31017647
- [Background] Pollack LA, Srinivasan A. Core elements of hospital antibiotic stewardship programs from the Centers for Disease Control and Prevention. Clin Infect Dis. 2014 Oct 15;59 Suppl 3(Suppl 3):S97-100. doi: 10.1093/cid/ciu542. PMID 25261548
- [Background] Rice LB. The Maxwell Finland Lecture: for the duration-rational antibiotic administration in an era of antimicrobial resistance and clostridium difficile. Clin Infect Dis. 2008 Feb 15;46(4):491-6. doi: 10.1086/526535. PMID 18194098
- [Background] Gupta K, Hooton TM, Naber KG, Wullt B, Colgan R, Miller LG, Moran GJ, Nicolle LE, Raz R, Schaeffer AJ, Soper DE; Infectious Diseases Society of America; European Society for Microbiology and Infectious Diseases. International clinical practice guidelines for the treatment of acute uncomplicated cystitis and pyelonephritis in women: A 2010 update by the Infectious Diseases Society of America and the European Society for Microbiology and Infectious Diseases. Clin Infect Dis. 2011 Mar 1;52(5):e103-20. doi: 10.1093/cid/ciq257. PMID 21292654
- [Background] Corona A, Bertolini G, Ricotta AM, Wilson A, Singer M. Variability of treatment duration for bacteraemia in the critically ill: a multinational survey. J Antimicrob Chemother. 2003 Nov;52(5):849-52. doi: 10.1093/jac/dkg447. Epub 2003 Sep 30. PMID 14519681
- [Background] Chotiprasitsakul D, Han JH, Cosgrove SE, Harris AD, Lautenbach E, Conley AT, Tolomeo P, Wise J, Tamma PD; Antibacterial Resistance Leadership Group. Comparing the Outcomes of Adults With Enterobacteriaceae Bacteremia Receiving Short-Course Versus Prolonged-Course Antibiotic Therapy in a Multicenter, Propensity Score-Matched Cohort. Clin Infect Dis. 2018 Jan 6;66(2):172-177. doi: 10.1093/cid/cix767. PMID 29190320
- [Background] Yahav D, Franceschini E, Koppel F, Turjeman A, Babich T, Bitterman R, Neuberger A, Ghanem-Zoubi N, Santoro A, Eliakim-Raz N, Pertzov B, Steinmetz T, Stern A, Dickstein Y, Maroun E, Zayyad H, Bishara J, Alon D, Edel Y, Goldberg E, Venturelli C, Mussini C, Leibovici L, Paul M; Bacteremia Duration Study Group. Seven Versus 14 Days of Antibiotic Therapy for Uncomplicated Gram-negative Bacteremia: A Noninferiority Randomized Controlled Trial. Clin Infect Dis. 2019 Sep 13;69(7):1091-1098. doi: 10.1093/cid/ciy1054. PMID 30535100
- [Background] Huttner A, Albrich WC, Bochud PY, Gayet-Ageron A, Rossel A, Dach EV, Harbarth S, Kaiser L. PIRATE project: point-of-care, informatics-based randomised controlled trial for decreasing overuse of antibiotic therapy in Gram-negative bacteraemia. BMJ Open. 2017 Jul 13;7(7):e017996. doi: 10.1136/bmjopen-2017-017996. PMID 28710229
- [Background] Schroeder S, Hochreiter M, Koehler T, Schweiger AM, Bein B, Keck FS, von Spiegel T. Procalcitonin (PCT)-guided algorithm reduces length of antibiotic treatment in surgical intensive care patients with severe sepsis: results of a prospective randomized study. Langenbecks Arch Surg. 2009 Mar;394(2):221-6. doi: 10.1007/s00423-008-0432-1. Epub 2008 Nov 26. PMID 19034493
- [Background] Nobre V, Harbarth S, Graf JD, Rohner P, Pugin J. Use of procalcitonin to shorten antibiotic treatment duration in septic patients: a randomized trial. Am J Respir Crit Care Med. 2008 Mar 1;177(5):498-505. doi: 10.1164/rccm.200708-1238OC. Epub 2007 Dec 20. PMID 18096708
- [Background] Corey GR, Stryjewski ME, Everts RJ. Short-course therapy for bloodstream infections in immunocompetent adults. Int J Antimicrob Agents. 2009;34 Suppl 4:S47-51. doi: 10.1016/S0924-8579(09)70567-9. PMID 19931818
- [Background] Havey TC, Fowler RA, Pinto R, Elligsen M, Daneman N. Duration of antibiotic therapy for critically ill patients with bloodstream infections: A retrospective cohort study. Can J Infect Dis Med Microbiol. 2013 Fall;24(3):129-37. doi: 10.1155/2013/141989. PMID 24421823
- [Background] Corona A, Wilson AP, Grassi M, Singer M. Prospective audit of bacteraemia management in a university hospital ICU using a general strategy of short-course monotherapy. J Antimicrob Chemother. 2004 Oct;54(4):809-17. doi: 10.1093/jac/dkh416. Epub 2004 Sep 16. PMID 15375106
- [Background] Cosgrove SE. The relationship between antimicrobial resistance and patient outcomes: mortality, length of hospital stay, and health care costs. Clin Infect Dis. 2006 Jan 15;42 Suppl 2:S82-9. doi: 10.1086/499406. PMID 16355321
- [Background] Maragakis LL, Perencevich EN, Cosgrove SE. Clinical and economic burden of antimicrobial resistance. Expert Rev Anti Infect Ther. 2008 Oct;6(5):751-63. doi: 10.1586/14787210.6.5.751. PMID 18847410
- [Background] Evans HL, Lefrak SN, Lyman J, Smith RL, Chong TW, McElearney ST, Schulman AR, Hughes MG, Raymond DP, Pruett TL, Sawyer RG. Cost of Gram-negative resistance. Crit Care Med. 2007 Jan;35(1):89-95. doi: 10.1097/01.CCM.0000251496.61520.75. PMID 17110877
- [Derived] Tingsgard S, Israelsen SB, Thorlacius-Ussing L, Frahm Kirk K, Lindegaard B, Johansen IS, Knudsen A, Lunding S, Ravn P, Ostergaard Andersen C, Benfield T. Short course antibiotic treatment of Gram-negative bacteraemia (GNB5): a study protocol for a randomised controlled trial. BMJ Open. 2023 May 8;13(5):e068606. doi: 10.1136/bmjopen-2022-068606. PMID 37156588

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT04291768/SAP_000.pdf